CLINICAL TRIAL: NCT05915039
Title: Usage of a Computer Assisted Learning (CAL) Module for Supplemental Re-training of BP Measurements by Doctor of Physical Therapy Students
Brief Title: Computer Assisted Learning (CAL) Module Use for Re-training of Blood Pressure Measurements by Physical Therapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-297
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure
Keywords: Physical Therapy; Education; Teaching

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized crossover design. Students enrolled in this study will undergo traditional blood pressure training. The students will be randomly divided into 2 groups (control and experimental). All students will undergo baseline testing 2 weeks after the class. At 48 hours before the 2 month timepoint, the experimental group will complete a CAL module entitled: "BP Measurement: Student Essentials". The control group will not undergo any retraining activities. All students will retest for accuracy, confidence, and knowledge. At the second 2 month mark, the control group will complete the CAL module and the experimental group will not. All students will retest for accuracy, confidence, and knowledge. All participants, the faculty teaching BP, and outcome assessors will be blinded from knowledge of groups throughout to reduce bias risk.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A faculty member without knowledge of the intervention and outcomes will randomize all subjects into 2 separate groups using random generated numbers from a computer software program:
  1. Control Group - Group "B" - Will not receive the CAL module training for the first retest session (T1), but will for T2.
  2. Experimental Group - Group "A" will complete the CAL module ahead of the first retest date (T1), but not for T2.
  Allocation of subjects to each group will be concealed in envelopes so that no other researcher knows who was assigned to a particular group (allocation concealment). The faculty member who performs the randomization and allocation will be the only researcher with knowledge of group allocation. This individual will open the envelopes and send the corresponding CAL module training link at the time points designated above. This faculty member is not involved in the class and has no knowledge of the outcomes or training provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This is the initial experimental group who will be exposed to the CAL module 48 hours before the first retesting period 2 months out from initial baseline measurement.
  Interventions: Other: Computer Assisted Learning (CAL) Module
- Group B (No Intervention): This is the initial control group who will not be exposed to the CAL module 48 hours before the first retesting period 2 months out from initial baseline measurement.

INTERVENTIONS:
Other: Computer Assisted Learning (CAL) Module — The students assigned to Group A will undergo interactive CAL module training by the American Medical Association which outlines how to properly measure blood pressure manually following the American Heart Association guidelines.
  Arms: Group A

SUMMARY:
The purpose of this study is to determine the effectiveness of a Computer Assisted Learning Module for supplemental blood pressure measurement retraining for doctor of physical therapy students.

ELIGIBILITY:
Inclusion Criteria:

1. Current student enrolled in the DPT program
2. Student is in good standing academically
3. Student is enrolled in the Clinical Foundation Skills course for the first time
4. Student provided informed consent to participate

Exclusion Criteria:

1. Student not enrolled in the DPT program
2. Student is taking the Clinical Skills Foundation course for the 2nd time
3. Student is not in good academic standing
4. Student did not provide informed consent to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of blood pressure measurements | Baseline to 4 months
  Pre-programmed manikin arms will be set to different blood pressure values. Students must correctly identify each of the pre-set blood pressure measurements
Confidence of blood pressure measurements | Baseline to 4 months
  A 5-point Likert scale survey to assess student confidence in different aspects of measuring blood pressure. The scale ranges from 1 to 5 with the following values: 1 - Not confident at all, 2 - Slightly confident, 3 - Moderately confident, 4 - Very confident, and 5 - extremely confident. A higher score indicates that the individual has higher levels of confidence for the reported item.
Blood pressure measurement knowledge quiz | Baseline to 4 months
  A knowledge quiz regarding the proper steps of blood pressure measurement as defined by the American Heart Association. This is a 15 question multiple choice quiz. The higher the score, the better the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Ickert, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmstrup M, Jensen B, Burkart R, Levis M. Using a novel assessment of procedural proficiency provides medical educators insight into blood pressure measurement. Int J Med Educ. 2016 Nov 19;7:375-381. doi: 10.5116/ijme.580b.2e4f. PMID 27864919
- [Background] Gordon CJ, Frotjold A, Fethney J, Green J, Hardy J, Maw M, Buckley T. The effectiveness of simulation-based blood pressure training in preregistration nursing students. Simul Healthc. 2013 Oct;8(5):335-40. doi: 10.1097/SIH.0b013e3182a15fa7. PMID 24061336
- [Background] Seybert AL, Barton CM. Simulation-based learning to teach blood pressure assessment to doctor of pharmacy students. Am J Pharm Educ. 2007 Jun 15;71(3):48. doi: 10.5688/aj710348. PMID 17619648
- [Background] Bland M, Ousey K. Preparing students to competently measure blood pressure in the real-world environment: a comparison between New Zealand and the United Kingdom. Nurse Educ Pract. 2012 Jan;12(1):28-35. doi: 10.1016/j.nepr.2011.04.009. Epub 2011 Jun 8. PMID 21641869
- [Background] Gazibara T, Rancic B, Maric G, Radovanovic S, Kisic-Tepavcevic D, Pekmezovic T. Medical students, do you know how to measure blood pressure correctly? Blood Press Monit. 2015 Feb;20(1):27-31. doi: 10.1097/MBP.0000000000000085. PMID 25243713
- [Background] Rakotz MK, Townsend RR, Yang J, Alpert BS, Heneghan KA, Wynia M, Wozniak GD. Medical students and measuring blood pressure: Results from the American Medical Association Blood Pressure Check Challenge. J Clin Hypertens (Greenwich). 2017 Jun;19(6):614-619. doi: 10.1111/jch.13018. Epub 2017 Apr 28. PMID 28452119
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Gonzalez-Lopez JJ, Gomez-Arnau Ramirez J, Torremocha Garcia R, Albelda Esteban S, Alio del Barrio J, Rodriguez-Artalejo F. Knowledge of correct blood pressure measurement procedures among medical and nursing students. Rev Esp Cardiol. 2009 May;62(5):568-71. doi: 10.1016/s1885-5857(09)71840-7. English, Spanish. PMID 19406072
- [Background] Crosley AM, Rose JR. Knowledge of accurate blood pressure measurement procedures in chiropractic students. J Chiropr Educ. 2013 Fall;27(2):152-7. doi: 10.7899/JCE-13-3. Epub 2013 Jun 27. PMID 23957320
- [Background] Ibiyemi O, Ogunbodede O, Gbolahan OO, Ogah OS. Knowledge and practices of blood pressure measurement among final year students, house officers, and resident dental surgeons in a dental hospital, South West Nigeria. Niger J Clin Pract. 2020 Jun;23(6):848-856. doi: 10.4103/njcp.njcp_416_19. PMID 32525122
- [Background] Rabbia F, Testa E, Rabbia S, Pratico S, Colasanto C, Montersino F, Berra E, Covella M, Fulcheri C, Di Monaco S, Buffolo F, Totaro S, Veglio F. Effectiveness of blood pressure educational and evaluation program for the improvement of measurement accuracy among nurses. High Blood Press Cardiovasc Prev. 2013 Jun;20(2):77-80. doi: 10.1007/s40292-013-0012-5. Epub 2013 May 8. PMID 23653174
- [Background] Leung GK, Nicholls JM. Effect of clinical context on simulator-based assessment of blood pressure taking - a pilot randomized study. Med Teach. 2014 Feb;36(2):177-9. doi: 10.3109/0142159X.2013.849328. Epub 2013 Oct 24. PMID 24156287
- [Background] Grim CM, Grim CE. A curriculum for the training and certification of blood pressure measurement for health care providers. Can J Cardiol. 1995 Nov;11 Suppl H:38H-42H. PMID 7489543